CLINICAL TRIAL: NCT06344065
Title: A Phase III, Single Center, Randomized, Blind, and Positive Control Clinical Trial to Evaluate the Immunogenicity and Safety of Diphtheria, Tetanus and Acellular Pertussis (Component) Combined Vaccine (Adsorbed) in 3-month-old Infants
Brief Title: Immunogenicity and Safety of Diphtheria, Tetanus, Pertussis (DTaP) Vaccine in 3-month-old Infants
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20220102C
Record Dates: First submitted 2024-03-11; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers
Keywords: DTaP
MeSH Terms: interventions — Tetanus Toxoid; Elements; Vaccines, Combined; Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DTaP vaccine (Experimental): Diphtheria, tetanus and acellular pertussis (component) combined vaccine (adsorbed), 0.5ml/vial, injection.
  Interventions: Biological: Diphtheria, tetanus and acellular pertussis (component) combined vaccine (adsorbed)
- Active comparator 1: DTaP vaccine (Active Comparator): Diphtheria, tetanus and acellular pertussis combined vaccine (adsorbed), 0.5ml/tube; injection.
  Interventions: Biological: Diphtheria, tetanus and acellular pertussis combined vaccine (adsorbed)
- Active comparator 2: DTaP-IPV//PRP-T vaccine (Active Comparator): Diphtheria, tetanus, pertussis (acellular, component), poliomyelitis (inactivated) vaccine (adsorbed) and Haemophilus influenzae type b conjugate vaccine, 0.5ml/tube; injection.
  Interventions: Biological: Diphtheria, tetanus, pertussis (acellular, component), poliomyelitis (inactivated) vaccine (adsorbed) and Haemophilus influenzae type b conjugate vaccine

INTERVENTIONS:
Biological: Diphtheria, tetanus and acellular pertussis (component) combined vaccine (adsorbed) — Three doses of basic immunization were administered at 3, 4, and 5 months of age, and one dose of booster immunization was administered at 18-24 months of age, for a total of four doses. The administration route for experimental vaccine is intramuscular injection of 0.5ml into the lateral deltoid muscle of the upper arm.
  Arms: DTaP vaccine
Biological: Diphtheria, tetanus and acellular pertussis combined vaccine (adsorbed) — Three doses of basic immunization were administered at 3, 4, and 5 months of age, and one dose of booster immunization was administered at 18-24 months of age, for a total of four doses. The administration route for active control vaccine 1 is intramuscular injection of 0.5ml into the lateral deltoid muscle of the upper arm.
  Arms: Active comparator 1: DTaP vaccine
Biological: Diphtheria, tetanus, pertussis (acellular, component), poliomyelitis (inactivated) vaccine (adsorbed) and Haemophilus influenzae type b conjugate vaccine — Three doses of basic immunization were administered at 3, 4, and 5 months of age, and one dose of booster immunization was administered at 18-24 months of age, for a total of four doses. The administration route for active control vaccine 2 is through intramuscular injection of 0.5ml into the anterolateral side of the thigh or the upper arm.
  Arms: Active comparator 2: DTaP-IPV//PRP-T vaccine

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of the DTaP in 3-month-old infants.

DETAILED DESCRIPTION:
This is a Phase III, Single Center, Randomized, Blind, and Positive Control Clinical Trial conducted in Guangxi Province, China. The purpose of this study is to evaluate the safety and immunogenicity of Diphtheria, Tetanus and Acellular Pertussis (Component) Combined Vaccine (Adsorbed) in 3-month-old infants. Expected to include 1584 3-month-old infants. Among them, 1056 infants were randomly assigned to the experimental group and active control group 1, and 528 infants were included in active control group 2. Select the top 200 subjects with study numbers from the experimental group as immunological persistence follow-up subset.

ELIGIBILITY:
Inclusion Criteria:

* Basic immune stage:

  1. 3-month-old infants who can provide valid identification documents;
  2. Infants should be born following a 37-42 weeks of pregnancy and have a birth weight that meets the standard (2500g ≤ body weight ≤ 4500g);
  3. The legal guardian of the subject voluntarily agrees to their child's participation in the trial and signs a written informed consent form;
  4. The legal guardian of the subject has the ability to understand the trial procedure and participate in all planned follow-up visits;
  5. Has not received a vaccine containing the active ingredients of pertussis, diphtheria, tetanus combined vaccine;
  6. Active control group 2 has not been vaccinated with any vaccine containing the active ingredients of poliomyelitis vaccine or haemophilus influenzae vaccine;
* Enhanced immunity stage:

  1. Infants and young children aged 18-24 months who have been enrolled in this clinical trial at the age of 3 months;
  2. Basic immunization has been completed in this clinical trial;
  3. According to the researcher's opinion, the subjects and their legal guardians are able to comply with the requirements of the clinical trial protocol.

Exclusion Criteria:

* Basic immune stage:

  1. Has a history of pertussis, diphtheria, or tetanus;
  2. Has any history of severe allergies to vaccination in the past;
  3. Allergy to any component of the experimental vaccine;
  4. Has a history or family history of epilepsy, convulsions, encephalopathy, mental illness;
  5. Individuals with thrombocytopenia, any coagulation dysfunction, or undergoing anticoagulant therapy that may cause contraindications for subcutaneous injection;
  6. Suffering from serious congenital malformations or serious diseases that may interfere with the conduct or completion of the trial including but not limited to: infant wheezing, Down syndrome, severe thalassemia, heart disease, liver disease, kidney disease, diabetes, hereditary allergies, Guillain Barre syndrome, severe skin diseases, congenital or acquired immune defects (repeated perianal abscess), etc;
  7. Has the history of severe abnormal production process, suffocation rescue, neurological damage, and current pathological jaundice;
  8. Suffering from infectious diseases with clinical or serological evidence, such as tuberculosis, hepatitis B, hepatitis C, or HIV infection confirmed by parents;
  9. Within 3 months before to enrollment, has received systemic corticosteroid treatment (any route of administration, ≥ 2mg/kg/day) for ≥ 14 days, such as prednisone, inhaled steroids such as budesonide, and fluticasone; Or being using other immunosuppressants such as cyclosporine, tacrolimus, etc. before enrollment;
  10. Within 3 months before enrollment，has received treatment with immunoglobulin and/or any blood products (except hepatitis B immunoglobulin) ;
  11. Participating in or planning to participate in clinical trials of other drugs in the near future;
  12. According to the researcher's judgment, there are any other factors that are not suitable for the subjects to participate in the clinical trial.
* Enhanced immunity stage:

  1. Newly discovered severe allergic history to any previous vaccination;
  2. Individuals with thrombocytopenia, any coagulation dysfunction, or undergoing anticoagulant therapy that may cause contraindications for subcutaneous injection;
  3. Suffering from serious congenital malformations or serious diseases that may interfere with the conduct or completion of the test, including but not limited to: infant wheezing, Down syndrome, severe thalassemia, heart disease, liver disease, kidney disease, diabetes, hereditary allergies, Guillain Barre syndrome, severe skin diseases, congenital or acquired immune defects (repeated perianal abscess), etc;
  4. After completing basic immunization, subjects were vaccinated with other vaccine containing the active ingredients of pertussis, diphtheria, tetanus combined vaccine before booster immunization;
  5. Participating in or planning to participate in clinical trials of other drugs in the near future;
  6. According to the researcher's judgment, there are any other factors that are not suitable for the subjects to participate in the clinical trial.

Ages: 3 Months to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1584 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-05-25 (Estimated); Study Completion 2028-12-25 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity results of experimental group and active control group (DTaP) | 30 days after basic immunization
  Positive conversion rate (4-fold increase) of antibodies against diphtheria (anti D) and tetanus (anti T)
Immunogenicity results of experimental group and active control group (DTaP-IPV//PRP-T) | 30 days after basic immunization
  Positive conversion rate (4-fold increase) of pertussis toxin antibody (anti PT), pertussis filamentous hemagglutinin antibody (anti FHA) antibodies
Immunogenicity results of experimental group | 30 days after basic immunization
  Positive conversion rate of pertussis adhesin antibody (anti PRN)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Du, Study Chair — Beijing Zhifei Lvzhu Biopharmaceutical Co., Ltd
Locations (1):
- Guangxi Zhuang Autonomous Region Center for Disease Control and Prevention, Nanning, Guangxi, China